CLINICAL TRIAL: NCT03483870
Title: Effect of Intravenous Granisetron on Incidence and Severity of Intrathecal Morphine Induced Pruritus in Elective Cesarean Section
Brief Title: Effect of Granisetron on Morphine Induced Pruritus in Cesarean Section
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rabab Ahmed Samy Anwer, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Granisetron in C.S
Record Dates: First submitted 2018-03-22; First posted 2018-03-30 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Pruritus
Keywords: Granisetron; Serum Serotonin; Morphine
MeSH Terms: conditions — Pruritus | interventions — Morphine; Saline Solution; Granisetron

STUDY DESIGN:
Intervention Model Description: comparison of the effect of intravenous granisetron with the effect of using placebo on morphine induced pruritus in parturients undergoing elective cesarean section under spinal anesthesia.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) The trial will be planned that neither the doctors (investigator) nor the parturients will be aware of the group allocation. The study drugs will be prepared by an anesthesiologist not involved in performing the intrathecal anesthesia, patient care or in data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morphine sulphate & Placebo (Placebo Comparator): 20 parturients under intrathecal anesthesia will receive 200 ug morphine sulphate intrathecally and 2 mL of normal saline 0.9% (placebo) IV injection preoperative.
  Interventions: Drug: Morphine Sulfate; Drug: Placebo
- Morphine sulphate & Granisetron (Active Comparator): 20 parturients under intrathecal anesthesia will receive 200 ug morphine sulphate intrathecally and 2 mL of 2 mg granisetron IV injection preoperative.
  Interventions: Drug: Morphine Sulfate; Drug: Granisetron

INTERVENTIONS:
Drug: Morphine Sulfate — 200 ug morphine sulphate will be injected intrathecally
Drug: Placebo — 2 mL of normal saline 0.9% IV injection
  Other Names: Normal saline 0.9%
  Arms: Morphine sulphate & Placebo
Drug: Granisetron — 2 mL of 2 mg granisetron IV injection
  Other Names: Kytril, Sancuso
  Arms: Morphine sulphate & Granisetron

SUMMARY:
Neuraxial anesthesia, which includes epidural anesthesia and intrathecal anesthesia, is a frequent anesthetic approach for caesarean delivery and other lower abdominal and lower limb anesthetic procedures. The addition of neuraxial morphine to local anesthetics provides an effective and prolonged postoperative analgesia. Neuraxial administration of morphine which is considered as a gold standard for analgesia has been associated with a frequent incidence of pruritus and postoperative nausea and vomiting.

The incidence of neuraxial opioid induced pruritus varies widely from 30% - 60% after orthopedic surgery with intrathecal morphine injection and from 60% - 100% in pregnant women after neuraxial opioid administration. Parturients appear to be the most susceptible to neuraxial opioid-induced pruritus which probably might be due to the interaction of estrogens with opioid receptors.

Although the exact mechanism of neuraxial opioid induced pruritus is unclear, the postulated mechanisms include the presence of an "itch center" in the central nervous system (CNS), medullary dorsal horn activation, antagonism of inhibitory transmitters, modulation of 5-hydroxytryptamine subtype 3 (5-HT3) or serotonergic pathways and the involvement of prostaglandins.

There is dense concentration of opioid receptors and 5-HT3 receptors in the dorsal part of the spinal cord and the nucleus of the spinal tract of the trigeminal nerve in the medulla. Activation of these receptors by neuraxial opioid administration or by circulating estrogen in parturients results in neuraxial opioid induced pruritus which is usually localized to the face, neck, or upper thorax. Nalbuphine, propofol and ondansetron have been used effectively in the treatment of pruritus associated with neuraxial morphine in surgical patients.

Granisetron is a potent and highly selective 5-HT3 receptor antagonist that has little or no affinity for other 5-HT receptors, or dopaminergic, adrenergic, benzodiazepine, histaminic, or opioid receptors. Its onset of action is 1-3 min, peak plasma level 30 min, plasma half-life is 4-6 h and duration of action up to 24 h. Its longer duration of action than that of ondansetron may coincide with the peak incidence of pruritus after intrathecal morphine (6-9 h). In contrast, other 5-HT3-receptor antagonists have affinities for various receptor-binding sites. For example, ondansetron has detectable binding to 5-HT1B, 5-HT1C, α1-adrenergic, and μ-opioid receptor sites. Although not proven, the binding of these agents to additional receptor subtypes other than their target receptor may underlie the inferior adverse event profile seen with ondansetron compared with granisetron.

DETAILED DESCRIPTION:
The study will be carried on 40 parturients scheduled for elective cesarean section (CS) under intrathecal anesthesia. They will be randomly allocated into two equal groups of 20 parturients each:

Group A: (placebo group) will receive 200 ug morphine sulphate will be injected intrathecally & 2 mL of normal saline 0.9%.

Group B: (treatment group) will receive 200 ug morphine sulphate will be injected intrathecally & 2 mL of 2 mg granisetron IV injection.

Preoperative assessment:

The day prior to surgery, all patients will undergo preanesthetic checkup including detailed history, thorough general, physical, systemic examination and weight of the patient. They will be kept NOP (nil per mouth) 6-8 hours for solids and 2 hours for water and clear fluids.

Preparation of the patients:

Written consent, coagulation profile, emergency resuscitation equipments including airway devices, advanced cardiac life support drugs. Parturients will be educated regarding the visual analogue scale (VAS).

Parturients in the holding area:

The patients will be positioned in the supine position, with uterine displacement to the left lateral side.

* Baseline monitoring readings of the maternal vital signs including Heart rate (HR), noninvasive systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), arterial oxygen saturation (SpO2) and respiratory rate (RR).
* Then IV cannula 18 G will be inserted into forearm vein and normal saline 0.9% solution 15 ml/kg will be infused for all women participating in the study over 20-30 minutes as a preload.
* The study drugs will be given 30 min before administration of intrathecal anesthesia.
* All patients will be premedicated with ranitidine 50 mg IV and then they will be transferred to the operating room.

Parturient in the operating room:

The previous monitoring data will be recorded again for the second time. Then subarachnoid block will be carried out under complete aseptic condition in the sitting position with the table in the horizontal level using 25 G pencil point spinal needle. Intrathecal block will be performed at the level of L 3-4 or L 4-5 vertebral interspaces; 12.5 mg (2.5 ml) of hyperbaric bupivacaine 0.5% and 200 ug morphine sulphate will be injected intrathecally at a rate of 1 ml/15 second after obtaining free flow of CSF. Immediately after end of injection of the drugs intrathecally, the parturient will be placed in the supine position with left lateral uterine displacement by putting a wedge under right hip (15ﹾ left-tilted supine position). All patients will receive supplemental oxygen 4 L/min via facemask until delivery of the baby. Sensory block will be assessed using loss of sensation in response to cold sensation (using ice cube). Surgery will start when the maximum height of sensory block reaches T6 or higher. Motor blockade will be assessed by modified Bromage scale (1 = unable to move feet or knees; 2 = able to move feet only; 3 = just able to move knees; 4 = full flexion of knees; 5 = no detectable weakness of hip flexion while supine; 6 = able to perform partial knee bend).

A third monitoring reading of the vital data will be taken immediately, 5 min and 10 min after spinal block and before the surgical operation (CS) starts.

Intraoperative assessment:

* After subarachnoid block parturients will be monitored for HR, NIBP, SpO2 and RR every 5 min till the end of the surgery. All parturients will be continuously monitored intraoperatively for any episodes of hypotension or bradycardia. Hypotension: defined as more than 20% decrease in maternal systolic blood pressure from the baseline. It will be treated with IV crystalloid fluid bolus and/or 3 mg IV ephedrine boluses when needed. Bradycardia defined as maternal heart rate < 60 beats/min. If occurred, it will be treated with IV atropine sulphate 0.5mg.
* After delivery of the baby, IV oxytocin 5 U will be administered slowly followed by an oxytocin infusion 0.03 U/mL at a rate of 200 mL/hr.

Study outcomes:

Primary outcome:

Incidence of pruritus during the first postoperative 24 hours.

Secondary outcomes:

1. Onset time of pruritus
2. Duration, location of pruritus and severity of pruritus according to the pruritus grading score The pruritus grading system (PGS) score for each patient is based on: distribution, frequency, severity of itch and quality of sleep.

   Pruritus Grading System

   Each patient's itch grade is calculated as the sum of the individual scores as:
   * Distribution:Solitary site 1, Multiple sites 2, Generalized 3
   * Frequency: Episodic 1, Frequent 3, Continuous 5
   * Severity: Rubbing 1, Scratching 1, Localized excoriations 3, Generalized excoriations 5
   * Sleep disturbance: Rare 0, Occasional 2, Frequent 4,Totally restless 6

   Mild grade: if total score is between 0 and 5.

   Moderate grade: if total score is between 6 and 11.

   Severe grade: if total score is between 12 and 19.

   The onset of pruritus will be assessed and recorded every 15 min for 4 hours along with the complaint by the patient. Pruritus scores will then be evaluated at 4, 8 and 24 hours post-surgery. For patients with pruritus who request treatment, antihistamines such as pheniramine maleate and μ-opioid receptor antagonists such as naloxone will be used depending upon the severity assessed by the clinician, if required.
3. Postoperative pain assessment, by a blinded Post-Anesthesia Care Unit (PACU) nurse using VAS at 6, 12, 18 and 24 hours after intrathecal morphine injection. Visual analog scale (Fig. 1) is a validated approach to pain measurement (Wood, 2004). The most common VAS consists of a 10-cm line with one end labeled "no pain" and the other end labeled "worst pain imaginable." The patient marks the line at the point that best describes the pain intensity. The length of the line to the patient's mark is measured and recorded in millimeters. The main theoretical advantage of the VAS is that it does not limit pain to 10 discrete levels of intensity, permitting a more detailed rating of pain.

   Rescue analgesia will be given in the form of perfalgan (paracetamol) 1 gm/ 6 h (max 4 gm per day) IV infusion and/or pethidine (meperidine) 1 mg/ kg IM when VAS is greater than 4.
4. Perioperative adverse events will be recorded, including nausea, vomiting (treated with 10 mg IV metoclopramide), intraoperative shortness of breath and respiratory depression (RR < 8 breaths/ min), and postoperative headache in the first 24 hours postoperatively.
5. Participants' satisfaction after end of the delivery: 1) not satisfied or 2) satisfied and willing to take the same medication and procedure in the future when indicated.

Serum serotonin measurment:

Two blood samples (2 mL each) will be withdrawn from each parturient. One sample will be withdrawn in the holding area before preload infusion and granisetron injection (basal reading for serum serotonin) and the other one will be withdrawn 6 hours after intrathecal morphine injection in both groups. Repeated freezing and thawing of the samples should be avoided. Hemolytic and especially lipemic serum samples should not be used with this assay. Storage: up to 6 hours at 2 - 8ºC; for longer periods (up to 6 months) at - 20 ºC.

Intended use and principle of the test: Enzyme Immunoassay for the quantitative determination of serotonin in serum. In the first step, serotonin is quantitatively acylated. The subsequent competitive ELISA kit uses the microtiter plate format. The antigen is bound to the solid phase of the microtiter plate. The acylated standards, controls and samples and the solid phase bound analyte compete for a fixed number of antiserum binding sites. After the system is in equilibrium, free antigen and free antigen-antiserum complexes are removed by washing. The antibody bound to the solid phase is detected by an anti-rabbit IgG-peroxidase conjugate using TMB as a substrate. The reaction is monitored at 450 nm.

Quantification of unknown samples is achieved by comparing their absorbance with a reference curve prepared with known standard concentrations. Expected reference values in serum: Males: 80 - 450 ng/ml and females: 40 - 400 ng/ml

ELIGIBILITY:
Inclusion Criteria:

* Parturients of American Society of Anesthesiologists (ASA) class I or II physical status.
* Age: 20-40 years.
* At term gestation (≥ 37 weeks) with a singleton uncomplicated pregnancy.
* Elective cesarean delivery under intrathecal anesthesia.

Exclusion Criteria:

* Parturient refusal.
* Significant organ dysfunctions (e.g., cardiac, respiratory, renal, or liver disorders).
* Morbid obesity (BMI >35).
* Parturients with known hypersensitivity to granisetron, morphine or amide local anesthetics.
* Parturients with pruritogenic systemic disease.
* A coexisting skin disorder or preexisting pregnancy induced pruritus.
* Parturients with any contraindication for intrathecal anesthesia, e.g. coagulopathy.
* Emergency cesarean section.
* Psychiatric disorders.
* Fetal abnormalities.
* Failed or unsatisfactory intrathecal block.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Incidence of pruritus during the first postoperative 24 hours. | 24 hours
  The effect of prophylactic intravenous (IV) administration of granisetron on incidence and severity of pruritus that occurs after intrathecal morphine in parturients undergoing cesarean section (CS).

SECONDARY OUTCOMES:
Onset time of pruritus | 24 hours
  Recording the time when itching began
The pruritus grading system (PGS) | 24 hours
  The pruritus grading system (PGS) score (Firas et al, 2012) for each patient is based on: distribution, frequency, severity of itch and quality of sleep.
  Each patient's itch grade is calculated as the sum of the individual scores as:
  Distribution:Solitary site 1, Multiple sites 2, Generalized 3
  Frequency: Episodic 1, Frequent 3, Continuous 5
  Severity: Rubbing 1, Scratching 1, Localized excoriations 3, Generalized excoriations 5
  Sleep disturbance: Rare 0, Occasional 2, Frequent 4,Totally restless 6
  Mild grade: if total score is between 0 and 5.
  Moderate grade: if total score is between 6 and 11.
  Severe grade: if total score is between 12 and 19.
Postoperative pain assessment | 24 hours
  Postoperative pain assessment, by a blinded Post-Anesthesia Care Unit (PACU) nurse using VAS at 6, 12, 18 and 24 hours after intrathecal morphine injection. Visual analog scale is a validated approach to pain measurement (Wood, 2004). The most common VAS consists of a 10-cm line with one end labeled "no pain" and the other end labeled "worst pain imaginable." The patient marks the line at the point that best describes the pain intensity. The length of the line to the patient's mark is measured and recorded in millimeters. The main theoretical advantage of the VAS is that it does not limit pain to 10 discrete levels of intensity, permitting a more detailed rating of pain.
  Rescue analgesia will be given in the form of perfalgan (paracetamol) 1 gm/ 6 h (max 4 gm per day) IV infusion and/or pethidine (meperidine) 1 mg/ kg IM when VAS is greater than 4.
Perioperative adverse events | 24 hours
  Nausea, vomiting, intraoperative shortness of breath and respiratory depression (RR < 8 breaths/ min), and postoperative headache in the first 24 hours postoperatively.
Participants' satisfaction after end of the delivery | 24 hours
  1) not satisfied or 2) satisfied and willing to take the same medication and procedure in the future when indicated.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kumar K, Singh SI. Neuraxial opioid-induced pruritus: An update. J Anaesthesiol Clin Pharmacol. 2013 Jul;29(3):303-7. doi: 10.4103/0970-9185.117045. PMID 24106351
- [Result] Dimitriou V, Voyagis GS. Opioid-induced pruritus: repeated vs single dose ondansetron administration in preventing pruritus after intrathecal morphine. Br J Anaesth. 1999 Nov;83(5):822-3. doi: 10.1093/bja/83.5.822. No abstract available. PMID 10690153
- [Result] Koju RB, Gurung BS, Dongol Y. Prophylactic administration of ondansetron in prevention of intrathecal morphine-induced pruritus and post-operative nausea and vomiting in patients undergoing caesarean section. BMC Anesthesiol. 2015 Feb 17;15:18. doi: 10.1186/1471-2253-15-18. PMID 25971957
- [Result] Szarvas S, Harmon D, Murphy D. Neuraxial opioid-induced pruritus: a review. J Clin Anesth. 2003 May;15(3):234-9. doi: 10.1016/s0952-8180(02)00501-9. PMID 12770663
- [Result] Blower P. A pharmacologic profile of oral granisetron (Kytril tablets). Semin Oncol. 1995 Aug;22(4 Suppl 10):3-5. No abstract available. PMID 7570052
- [Result] Breen TW, Shapiro T, Glass B, Foster-Payne D, Oriol NE. Epidural anesthesia for labor in an ambulatory patient. Anesth Analg. 1993 Nov;77(5):919-24. doi: 10.1213/00000539-199311000-00008. PMID 8214727
- [Result] Reich A, Szepietowski JC. Opioid-induced pruritus: an update. Clin Exp Dermatol. 2010 Jan;35(1):2-6. doi: 10.1111/j.1365-2230.2009.03463.x. Epub 2009 Jul 29. PMID 19663845
- [Result] Charuluxananan S, Kyokong O, Somboonviboon W, Narasethakamol A, Promlok P. Nalbuphine versus ondansetron for prevention of intrathecal morphine-induced pruritus after cesarean delivery. Anesth Analg. 2003 Jun;96(6):1789-1793. doi: 10.1213/01.ANE.0000066015.21364.7D. PMID 12761013
- [Result] Wood S. Factors influencing the selection of appropriate pain assessment tools. Nurs Times. 2004 Aug 31-Sep 6;100(35):42-7. PMID 15471273
- [Result] van Wijngaarden I, Tulp MT, Soudijn W. The concept of selectivity in 5-HT receptor research. Eur J Pharmacol. 1990 Jun 12;188(6):301-12. doi: 10.1016/0922-4106(90)90190-9. PMID 2164935
- [Result] Perez EA, Hesketh P, Sandbach J, Reeves J, Chawla S, Markman M, Hainsworth J, Bushnell W, Friedman C. Comparison of single-dose oral granisetron versus intravenous ondansetron in the prevention of nausea and vomiting induced by moderately emetogenic chemotherapy: a multicenter, double-blind, randomized parallel study. J Clin Oncol. 1998 Feb;16(2):754-60. doi: 10.1200/JCO.1998.16.2.754. PMID 9469367
- [Result] Slappendel R, Weber EW, Benraad B, van Limbeek J, Dirksen R. Itching after intrathecal morphine. Incidence and treatment. Eur J Anaesthesiol. 2000 Oct;17(10):616-21. doi: 10.1046/j.1365-2346.2000.00727.x. PMID 11050519
- See also: Using Pruritus Grading System for Measurement of Pruritus in Patients with Diseases Associated with Itch — http://journals.ju.edu.jo/JMJ/article/view/3023/5700